CLINICAL TRIAL: NCT00491166
Title: A Single-Center, Investigator-Sponsored Pilot Study to Assess Safety and Biologic Activity of Bromfenac Ophthalmic Solution, 0.09%, in Subjects With Diffuse DME Refractory to Laser
Brief Title: Safety Study of Bromfenac Ophthalmic Solution in Subjects With Diffuse Diabetic Macular Edema (DME) Refractory to Laser
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ophthalmic Consultants of Boston (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X-DME-001
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; bromfenac ophthalmic solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bromfenac ophthalmic solution

SUMMARY:
This is an investigator-sponsored trial (IST), an open-label pilot study, assessing the safety and biologic activity of bromfenac in subjects with diffuse DME refractory to laser.

DETAILED DESCRIPTION:
Ten subjects will be enrolled in this study, which will be conducted at Ophthalmic Consultants of Boston, Boston, MA. All subjects must be diagnosed with diffuse DME that is either refractory to laser photocoagulation or in patients who have refused laser.

Consented subjects will be screened to determine eligibility. Eligibility will be determined by the Investigator, a retinal specialist. Only one eye will be chosen as the "study eye." Only the study eye will receive bromfenac drops during the study.

Eligible subjects will self-administer bromfenac two times per day (BID) for three months (treatment period). Subjects will have monthly examinations during the treatment period, followed by follow up visits at Month 4 and Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Center-involved macular edema secondary to diabetes mellitus

Exclusion Criteria:

* Study eye with edema amenable to focal laser
* Treatment with laser, intraocular steroids, and anti-VEGF agents within 90 days
* Current eye infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
The mean change in visual acuity and central retinal thickness from baseline to month 3,and the incidence and severity of ocular adverse events and other adverse events. | Baseline to month 3

SECONDARY OUTCOMES:
Changes in retinal leakage as determined by fluorescein angiography | Baseline to month 3

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States